CLINICAL TRIAL: NCT00944827
Title: The Effects of Catechin Supplementation (Green Tea Extract), in Combination With the Classic Treatment for the Reduction of Hypercholesterolemia (Statin Therapy) on the Treatment's Effectiveness and in the Reduction of Classic Side Effects.
Brief Title: Combination Treatment With Green Tea Extract and Statins in Patients With Hypercholesterolemia
Acronym: GTE-Stat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Greek Ministry of Development (Other Government); General Hospital of Trikala, Dept of Internal Medicine (Unknown); University General Hospital of Larissa, Dept of Medicine (Unknown)
Responsible Party: Dr. Giorgos K. Sakkas, CERETETH - PerfoTech - ClinLab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 3-22/846/06-2007; 22/08-06-2007; no3/10-01-2007; 846/22/15-06-2007
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2009-07

CONDITIONS: Hypercholesterolemia
Keywords: Green Tea Extract; Catechins; Statin; atorvastatin; body composition; visceral fat; steatosis; oxidative stress; quality of life; OGTT; OGIS; ISI matsuda
MeSH Terms: conditions — Hypercholesterolemia; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GTE (Experimental): The experimental group will receive 20 mg atorvastatin (Lipitor) daily and 600 mg. of pure catechin in capsules
  Interventions: Dietary Supplement: Green Tea Extract - Catechins
- CON (Placebo Comparator): The control group will receive 20 mg atorvastatin (Lipitor) and Placebo in identical capsules containing 600 mg placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Green Tea Extract - Catechins — Combination treatment with 20 mg atorvastatin and 600mg green tea extract, daily for 12 weeks
  Arms: GTE
Dietary Supplement: Placebo — Combination treatment with 20 mg atorvastatin and 600mg placebo, daily for 12 weeks
  Arms: CON

SUMMARY:
There is a positive correlation between serum's cholesterol levels and death from cardiovascular disease, especially coronary artery disease. The reduction of plasma lipids levels is one of the main goals of prevention. Research has shown that green tea has beneficial effects on health due to the polyphenolic substances (catechins) that it contains. Studies have shown that prolonged consumption of polyphenols has a positive effect on factors related to cardiovascular risk such as obesity, dislipidemia and various indicators of oxidative stress.

The aim of this study was to examine the possible effects of catechin supplementation, in combination with the classic treatment for the reduction of hypercholesterolemia, statin therapy, on the treatment's effectiveness and in the reduction of classic side effects.

DETAILED DESCRIPTION:
This is a randomized, double - blind placebo controlled trial. The patients will be divided randomly in two groups; one group will receive statin and catechin, while the other statin and placebo for 12 weeks. The experimental group will receive 20 mg atorvastatin (Lipitor) daily and 600 mg of catechin in capsules, while the control group will receive 20 mg atorvastatin (Lipitor) and Placebo in identical capsules of 600 mg for the same time period.

The patients will undergo biochemical evaluation in which the serum lipids, the levels of oxidative stress and the antioxidant capacity will be assessed. Body composition will be calculated with anthropometric measurements, while the levels of visceral fat, the subcutaneous fat, as well as the level of liver fat infiltration will be examined with the use of computed tomography images. Factors related to the patients' quality of life will be assessed by a series of questionnaires.

The investigators hypothesized that the combination treatment with statin and green tea extract (catechins)will improve in a greater extent the lipidemic profile, increase antioxidant capacity, reducing significantly visceral fat and intrahepatic lipids content.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol >200mg/dl, or LDL >160 mg/dl

Exclusion Criteria:

* normal lipidemic profile, on statin medication, diabetes mellitus, liver disease, severe hypertension, pregnancy, or severe side effects after 4 weeks of treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Reduction in Total CHO and LDH | 12 wks

SECONDARY OUTCOMES:
lipids profile, body composition, visceral adiposity, Redox status, glucose disposal, Insulin sensitivity index, liver fat infiltration, quality of life parameters | 12 wks

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos K Sakkas, PhD, Principal Investigator — UTH - CERETETH; Christina Karatzaferi, PhD, Principal Investigator — University of Thessaly
Locations (1):
- General Hospital of Trikala, Trikala, Thessaly, Greece